CLINICAL TRIAL: NCT01464944
Title: A Randomized, Double-blind, Double-dummy, Single-dose, Parallel Group, Multicenter Study to Compare the Antipyretic Efficacy of Acetylsalicy-lic Acid 500 mg and 1,000 mg (2 x 500 mg) and Paracetamol 500 mg and 1,000 mg (2 x 500 mg) With Placebo in Patients With Acute Febrile Upper Respiratory Tract Infections Suspected to be of Viral Origin.
Brief Title: Placebo and Active Controlled Study to Compare the Antipyretic Efficacy of Aspirin® in Patients With Acute Febrile Upper Respiratory Tract Infections Suspected to be of Viral Origin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11202
Record Dates: First submitted 2011-05-17; First posted 2011-11-04 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Respiratory Tract Infections; Fever
Keywords: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections; Fever | interventions — Aspirin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 2 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Arm 3 (Active Comparator)
  Interventions: Drug: Paracetamol
- Arm 4 (Active Comparator)
  Interventions: Drug: Paracetamol
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Acetylsalicylic acid 500 mg orally, single dose, 1 tablet; in addition, 1 Placebo tablet of Acetylsalicylic acid, and 2 Placebo tablets of Paracetamol
  Arms: Arm 1
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Acetylsalicylic acid 2 x 500 mg orally, single dose, 2 tablets; in addition, 2 Placebo tablets of Paracetamol
  Arms: Arm 2
Drug: Paracetamol — Paracetamol 500 mg orally, single dose, 1 tablet; in addition, 1 Placebo tablet of Paracetamol, and 2 Placebo tablets of Acetylsalicylic Acid
  Arms: Arm 3
Drug: Paracetamol — Paracetamol 2 x 500 mg orally, single dose, 2 tablets; in addition, 2 Placebo tablets of Acetylsalicylic Acid
  Arms: Arm 4
Drug: Placebo — 2 Placebo tablets of Acetylsalicylic Acid, and 2 Placebo tablets of Paracetamol, orally, single dose
  Arms: Arm 5

SUMMARY:
This study is addressed to patients suffering from an acute febrile upper respiratory tract infection suspected to be of viral origin. The purpose of this study is to determine the antipyretic efficacy (reduction of fever by lowering the body temperature from a raised state) of Aspirin in doses of 500 and 1000 mg (study medication) compared to the one of Paracetamol in doses of 500 and 1000 mg (comparator medication) as well as the one of Placebo (comparator medication without an active substance). Despite of its common use for fever treatment, the scientific data in adults which support the antipyretic efficacy of Aspirin are sparse. Therefore, the purpose of this study is to collect such data.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patients 18 to 65 years of age
* Acute uncomplicated febrile URTI suspected to be of viral origin and present not more than 5 days
* Symptoms of a viral URTI
* Oral temperature >/= 38.5 °C to </= 40°C

Exclusion Criteria:

* Patients with physical findings consistent with the diagnosis of pneumonia, otitis media, bacterial sinusitis or any other bacterial infection of the respiratory tract requiring antibiotics or other therapeutic intervention by a physician
* Current antibiotic treatment or pre-treatment with antibiotic agents during the last week
* History or presence of asthma or hypersensitivity to ASA, salicylates, paracetamol, or other non-steroidal anti-inflammatory drugs; peptic ulceration or gastric bleeding; hemorrhagic diathesis; hepatic and/or renal dysfunction; Gilbert's disease; Quincke's edema
* Any other acute or chronic disease which in the opinion f the investigator could interfere with the patient's health and well-being during the conduct of the study or which could interfere with the evaluation of data generated from this subject
* Any conditions possibly interfering with the gastro-intestinal absorption of the study medication
* Pregnant or lactating women. All women of childbearing age were to undergo a pregnancy test before start of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2003-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the orally measured change of body temparature from baseline over a period of 0 - 4 hours post dose. | Up to 4 hours post dose

SECONDARY OUTCOMES:
Maximum temperature difference between baseline and the lowest measured temperature | Up to 4 hours post dose
Time to reach the maximum temperature difference | Up to 4 hours post dose
Intensity of Upper Respiratory Tract Infection symptoms | 0, 2, 4, and 6 hours post dose
Safety - assessment of adverse events | Up to 7 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Moscow, Russia
- Ukraine (2):
  - Kiev
  - Luhansk